CLINICAL TRIAL: NCT06426316
Title: Immune System, Inflammation, Migraine - The Role of Cytokines and Regulatory T Lymphocytes in Migraine Pathophysiology
Brief Title: The Role of Cytokines and Regulatory T Lymphocytes in Migraine Pathophysiology.
Acronym: SIIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2023 STUCHFIELD; 2023-A01503-42 (Other: ANSM)
Record Dates: First submitted 2024-04-30; First posted 2024-05-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-06

CONDITIONS: Migraine Disorders; Pain; Autoimmune Diseases; Multiple Sclerosis; Endometriosis; Rheumatoid Arthritis; Crohn Disease; Lupus Erythematosus
Keywords: Migraine Disorders; Pain; Cytokines; Regulatory T cell
MeSH Terms: conditions — Migraine Disorders; Pain; Autoimmune Diseases; Multiple Sclerosis; Endometriosis; Arthritis, Rheumatoid; Crohn Disease | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Migraine - no autoimmune/inflammatory disease (Experimental): Migraine - no autoimmune/inflammatory disease group
  Interventions: Biological: Blood test
- No migraine - no autoimmune/inflammatory disease (Experimental): No migraine - no autoimmune/inflammatory disease group
  Interventions: Biological: Blood test
- No migraine - autoimmune/inflammatory disease (MS, RA, CD, SLE, T1DM, endometriosis) (Experimental): No migraine - autoimmune/inflammatory disease (MS, RA, CD, SLE, T1DM, endometriosis) group
  Interventions: Biological: Blood test
- Migraine - autoimmune/inflammatory disease (MS, RA, CD, SLE, T1DM, endometriosis) (Experimental): Migraine - autoimmune/inflammatory disease (MS, RA, CD, SLE, T1DM, endometriosis) group
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — 1 blood test of maximum 40 millilitres per patient

SUMMARY:
Migraine is a frequent and debilitating neurologic disorder. It is more frequent in women, and more prevalent in patients with autoimmune and/or inflammatory diseases such as multiple sclerosis (MS), rheumatoid arthritis (RA), Crohn's disease (CD), systemic lupus erythematosus (SLE) and endometriosis, whereas patients with long standing type 1 diabetes mellitus (T1DM) - an autoimmune but non inflammatory disease - seem to be less affected compared to the general population. Despite new migraine prevention treatments, a large number of patients remain unresponsive to currently available anti-migraine therapy and migraine pathophysiology remains unclear. Several peptides (calcitonin gene-related peptide (CGRP), pituitary adenylate cyclase activating peptide-38 (PACAP-38), vasoactive intestinal polypeptide (VIP)) and hormones (estrogens, prolactin) and the immune system play an important role in migraine pathophysiology. Among T lymphocytes, regulatory T (Treg) cells suppress inflammation. Studies have evidenced higher levels of inflammatory molecules (cytokines) in migraine patients and have suggested decreased proportions of Treg cells in migraine, as well as in MS, RA, CD and SLE, whereas inflammation declines and Treg levels seem increased in long-standing T1DM. Inflammation, which participates in migraine pain, seems to be a common factor for migraine and these diseases. However, these studies display conflicting results and further investigation is required to better understand the mechanisms behind migraine.

In this study, the investigators will compare Treg levels, as well as identify Treg subpopulations and measure cytokine levels in migraine and migraine-free participants with and without an autoimmune/inflammatory disorder (MS, RA, CD, SLE, T1DM and endometriosis).

DETAILED DESCRIPTION:
Migraine is the 6th most frequent disease (14% of the population) and the second leading cause of disability worldwide. From puberty and onward, migraine is 2 to 3 times more frequent in women, which also suffer from more severe attacks. Migraine is also up to twice as prevalent in patients suffering from autoimmune or inflammatory diseases such as multiple sclerosis (MS), rheumatoid arthritis (RA), Crohn disease (CD), systemic lupus erythematosus (SLE) and endometriosis, whereas patients with long standing type 1 diabetes mellitus (T1DM) - an autoimmune but non inflammatory disease - seem to be less affected compared to the general population.

Despite the identification of the role of peptides such as CGRP in migraine pathophysiology and the development of targetted anti-CGRP treatments, many patients remain unresponsive and the mechanisms behind migraine are still unclear.

The trigemino-vascular system is involved in the perception of migraine pain. Migraine occurs with trigemino-cervical neuron sensitization, leading to peptide secretion (such as CGRP, PACAP-38 and VIP), which induce neurogenic inflammation that is responsible for vasodilation, capillary leakage, oedema and further sensitization of the trigemino-vascular system, leading to amplified perception of migraine pain. CGRP, PACAP-38 and VIP infusions all induce migraine attacks in migraine patients, and only mild or no headache in healthy volunteers.

Sex hormones, prolactin and insulin are also involved in migraine pathophysiology, and the immune system, through cytokine production and immune cell dysregulations seems to also play a role in the pathogenesis of migraine. Both are closely related as sex hormone levels may have an influence on the levels of certain immune cell subtypes. Several pro-inflammatory cytokines (tumor necrosis factor (TNF)-alpha, interferon (IFN)-gamma and interleukin (IL)-6) were shown to be elevated in migraine patients but also inflammatory diseases such as MS and endometriosis compared to controls and are associated with migraine pathophysiology. Inflammation seems to be a common factor for migraine and these diseases. However, these studies provide conflicting results and further investigation is needed to better understand the role of inflammation in migraine pathophysiology.

Among T lymphocytes, regulatory T (Treg) cells regulate inflammation by suppressing effector T cells through several suppressive mechanisms such as IL-10 secretion or the hydrolysis of pro-inflammatory and nociceptive adenosine triphosphate (ATP) into anti-inflammatory and anti-nociceptive adenosine by cluster of differentiation (CD) 39 and 73 enzymes on the Treg cell surface. Recent studies have suggested decreased Treg proportions in migraine patients, particularly CD 39 and CD 73-positive Treg cells, whereas Treg cells were shown to be increased in T1DM patients. This suggests the role of Treg cells in migraine, but further studies are needed.

In this study, the investigators aim to compare Treg levels, as well as identify Treg subpopulations and measure cytokine levels in migraine and migraine-free participants with and without an autoimmune/inflammatory disorder (MS, RA, CD, SLE, T1DM and endometriosis). This will provide better understanding of migraine pathophysiology and lead to the development of targeted and personalized treatment strategies, according to the immune pain profile and associated inflammatory diseases of migraine patients.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 - 50 years of age
* at least 50 kg
* autoimmune/inflammatory disease groups : with a diagnosis of multiple sclerosis, systemic lupus erythematous, rheumatoid arthritis, Crohn's disease, type 1 diabetes or endometriosis
* migraine group : with a diagnosis of migraine with at least 4 headache days per month

Exclusion Criteria:

* BMI < or = 17 ou > or = 30kg/m²
* type 2 diabetes, immune deficit, other chronic autoimmune or inflammatory disease
* non-migraine headache, except for tension type headache of less than 4 days/month
* pregnancy, delivery, miscarriage, breast-feeding, participation in a medically assisted human reproduction program (ovary stimulation/hormone therapy) < 3 months before blood sampling
* Menopause, hysterectomy, or bilateral oophorectomy
* Hormone therapy (besides contraception and treatment of endometriosis)
* bone marrow or solid organ transplant
* guardianship, curatorship, safeguard of justice or deprivation of liberty
* for patients : diagnosis of several autoimmune or inflammatory diseases
* for controls : diagnosis of an autoimmune or inflammatory disease
* for non-migraine participants : migraine

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 396 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Treg cell levels in cell/microliter (cell/µL) and percentage (%) of white blood cells | Once, at inclusion
  To measure Treg cell levels in migraine and migraine-free participants, with and without autoimmune/inflammatory diseases (MS, RA, CD, SLE, endometriosis, T1DM) using flow cytometry

SECONDARY OUTCOMES:
Cytokine levels in picogram per milliliter (pg/mL) | Once, at inclusion
  To measure cytokine levels (interleukin 1a and b, interleukin 2, interleukin 6, interleukin 10, interleukin 12, interleukin 17, interleukin 18, interleukin 21, interleukin 22, interleukin 23, interleukin 33, interleukin 35, interleukin 36b, interleukin 37, interleukin 38, tumor necrosis factor a, interferon g, transforming growth factor b, interleukin 1ra, C-C motif ligand 20) using a LUMINEX method
Impact of hormones (progesterone, estrogen, testosterone, follicle stimulating hormone (FSH), luteinizing hormone (LH), insulin and prolactin) levels on levels of Treg cells | Once, at inclusion
  To determine the impact of hormones on Treg cell levels
Impact of hormones (progesterone, estrogen, testosterone, follicle stimulating hormone (FSH), luteinizing hormone (LH), insulin and prolactin) levels on levels of cytokines | Once, at inclusion
  To determine the impact of hormones on cytokine levels
Impact of neuropeptides (calcitonin gene-related peptide (CGRP), vasoactive intestinal polypeptide (VIP), pituitary adenylate cyclase-activating polypeptide (PACAP) on Treg cell levels | Once, at inclusion
  To determine the impact of neuropeptides on Treg cell levels
Impact of neuropeptides (calcitonin gene-related peptide (CGRP), vasoactive intestinal polypeptide (VIP), pituitary adenylate cyclase-activating polypeptide (PACAP) on cytokine levels | Once, at inclusion
  To determine the impact of neuropeptides on cytokine levels

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MOISSET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand - Service de Neurologie, Clermont-Ferrand, AURA, France

REFERENCES:
- [Background] Chan HS, DeBoer G, Haddad G, Gallie BL, Ling V. Multidrug resistance in pediatric malignancies. Hematol Oncol Clin North Am. 1995 Apr;9(2):275-318. PMID 7642465
- [Background] Supabphol R, Stewart PJ. Influence of the carrier on the intrinsic rate of dissolution of diazepam in interactive mixtures. J Pharm Pharmacol. 1996 Dec;48(12):1249-55. doi: 10.1111/j.2042-7158.1996.tb03931.x. PMID 9004186
- [Background] Ashina M. Migraine. N Engl J Med. 2020 Nov 5;383(19):1866-1876. doi: 10.1056/NEJMra1915327. No abstract available. PMID 33211930
- [Background] Takami H, Miyaji S, Koudaira H, Kodaira S, Sugawara I. [Role in mucosal ornithine decarboxylase activity during dimethylhydrazine-induced colonic carcinogenesis in the rat]. Gan To Kagaku Ryoho. 1993 Aug;20(10):1405-7. No abstract available. Japanese. PMID 8346940
- [Background] Al-Karagholi MA, Kalatharan V, Ghanizada H, Gram C, Dussor G, Ashina M. Prolactin in headache and migraine: A systematic review of clinical studies. Cephalalgia. 2023 Feb;43(2):3331024221136286. doi: 10.1177/03331024221136286. PMID 36718026
- [Background] Coble BI, Briheim G, Dahlgren C, Molin L. Function of exudate neutrophils from skin in psoriasis. Int Arch Allergy Appl Immunol. 1988;85(4):398-403. doi: 10.1159/000234541. PMID 3356472
- [Background] Stevensjc, Marks LE, Gagge AP. The quantitative assessment of thermal discomfort. Environ Res. 1969 Apr;2(3):149-65. doi: 10.1016/0013-9351(69)90035-8. No abstract available. PMID 5788906
- [Background] Watkins LR, Maier SF. Glia: a novel drug discovery target for clinical pain. Nat Rev Drug Discov. 2003 Dec;2(12):973-85. doi: 10.1038/nrd1251. No abstract available. PMID 14654796
- [Background] Perini F, D'Andrea G, Galloni E, Pignatelli F, Billo G, Alba S, Bussone G, Toso V. Plasma cytokine levels in migraineurs and controls. Headache. 2005 Jul-Aug;45(7):926-31. doi: 10.1111/j.1526-4610.2005.05135.x. PMID 15985111
- [Background] Vignali DA, Collison LW, Workman CJ. How regulatory T cells work. Nat Rev Immunol. 2008 Jul;8(7):523-32. doi: 10.1038/nri2343. PMID 18566595
- [Background] Arumugam M, Parthasarathy V. Reduction of CD4(+)CD25(+) regulatory T-cells in migraine: Is migraine an autoimmune disorder? J Neuroimmunol. 2016 Jan 15;290:54-9. doi: 10.1016/j.jneuroim.2015.11.015. Epub 2015 Nov 28. PMID 26711570
- [Background] Faraji F, Shojapour M, Farahani I, Ganji A, Mosayebi G. Reduced regulatory T lymphocytes in migraine patients. Neurol Res. 2021 Aug;43(8):677-682. doi: 10.1080/01616412.2021.1915077. Epub 2021 Apr 14. PMID 33853506
- [Background] Okimura H, Tanaka Y, Fujii M, Shimura K, Maeda E, Ito F, Khan KN, Nakamura Y, Mori T, Kitawaki J. Changes in the proportion of regulatory T cell subpopulations during menstrual cycle and early pregnancy. Am J Reprod Immunol. 2022 Dec;88(6):e13636. doi: 10.1111/aji.13636. Epub 2022 Oct 21. PMID 36217280
- [Background] Moisset X, Bommelaer G, Boube M, Ouchchane L, Goutte M, Dapoigny M, Dallel R, Guttmann A, Clavelou P, Buisson A. Migraine prevalence in inflammatory bowel disease patients: A tertiary-care centre cross-sectional study. Eur J Pain. 2017 Oct;21(9):1550-1560. doi: 10.1002/ejp.1056. Epub 2017 May 16. PMID 28508514
- [Background] Moisset X, Giraud P, Dallel R. Migraine in multiple sclerosis and other chronic inflammatory diseases. Rev Neurol (Paris). 2021 Sep;177(7):816-820. doi: 10.1016/j.neurol.2021.07.005. Epub 2021 Jul 27. PMID 34325914
- [Background] Yang MH, Wang PH, Wang SJ, Sun WZ, Oyang YJ, Fuh JL. Women with endometriosis are more likely to suffer from migraines: a population-based study. PLoS One. 2012;7(3):e33941. doi: 10.1371/journal.pone.0033941. Epub 2012 Mar 19. PMID 22442736
- [Background] Hagen K, Asvold BO, Midthjell K, Stovner LJ, Zwart JA, Linde M. Inverse relationship between type 1 diabetes mellitus and migraine. Data from the Nord-Trondelag Health Surveys 1995-1997 and 2006-2008. Cephalalgia. 2018 Mar;38(3):417-426. doi: 10.1177/0333102417690488. Epub 2017 Jan 23. PMID 28114807
- [Background] Malutan AM, Drugan T, Costin N, Ciortea R, Bucuri C, Rada MP, Mihu D. Pro-inflammatory cytokines for evaluation of inflammatory status in endometriosis. Cent Eur J Immunol. 2015;40(1):96-102. doi: 10.5114/ceji.2015.50840. Epub 2015 Apr 22. PMID 26155190
- [Background] Gobel K, Ruck T, Meuth SG. Cytokine signaling in multiple sclerosis: Lost in translation. Mult Scler. 2018 Apr;24(4):432-439. doi: 10.1177/1352458518763094. Epub 2018 Mar 7. PMID 29512406
- [Background] Shi JL, Zheng ZM, Chen M, Shen HH, Li MQ, Shao J. IL-17: an important pathogenic factor in endometriosis. Int J Med Sci. 2022 Apr 11;19(4):769-778. doi: 10.7150/ijms.71972. eCollection 2022. PMID 35582411
- [Background] Viisanen T, Gazali AM, Ihantola EL, Ekman I, Nanto-Salonen K, Veijola R, Toppari J, Knip M, Ilonen J, Kinnunen T. FOXP3+ Regulatory T Cell Compartment Is Altered in Children With Newly Diagnosed Type 1 Diabetes but Not in Autoantibody-Positive at-Risk Children. Front Immunol. 2019 Jan 22;10:19. doi: 10.3389/fimmu.2019.00019. eCollection 2019. PMID 30723474